CLINICAL TRIAL: NCT03973268
Title: The Mechanism of Action Underlying Ketamine's Antidepressant Effects: An Investigation of the AMPA Throughput Theory in Patients With Treatment-Resistant Major Depression
Brief Title: Mechanism of Action Underlying Ketamine's Antidepressant Effects: The AMPA Throughput Theory in Patients With Treatment-Resistant Major Depression
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 190107; 19-M-0107
Record Dates: First submitted 2019-06-01; First posted 2019-06-04 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12-08

CONDITIONS: Depression; Major Depressive Disorder; Major Depression
Keywords: Biomarker; AMPA Antagonist; Magnetoencephalography; Neuropharmacology; Neurobiology
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- 1 (Experimental): Individuals in Arm 1 will receive double-blinded perampanel and open-label ketamine on the first day, then double-blinded perampanel on the second day.
  Interventions: Device: Arm 1, 2, 3 device interventions; Drug: Arm 1, 2, 3 drug Interventions; Drug: Arm 1 and 2 Interventions
- 2 (Experimental): Individuals in Arm 2 will receive double-blinded placebo and open-label ketamine on the first day, then double-blinded perampanel on the second day.
  Interventions: Device: Arm 1, 2, 3 device interventions; Other: Arm 2 Interventions; Drug: Arm 1, 2, 3 drug Interventions; Drug: Arm 1 and 2 Interventions
- 3 (Experimental): Individuals in Arm 3 will receive double-blinded placebo and open-label ketamine on the first day, then double-blinded placebo on the second day.
  Interventions: Device: Arm 1, 2, 3 device interventions; Drug: Arm 1 and 2 Interventions

INTERVENTIONS:
Device: Arm 1, 2, 3 device interventions — MagPro 100 TMS Therapy System
Other: Arm 2 Interventions — Placebo
  Arms: 2
Drug: Arm 1, 2, 3 drug Interventions — Ketamine
  Arms: 1; 2
Drug: Arm 1 and 2 Interventions — Perampanel

SUMMARY:
Background:

Most drugs that treat mood disorders take a long time to work. Ketamine works within hours. A dose can last for a week or more. Certain receptors in the brain might help ketamine work. A drug that blocks these receptors might affect how it works.

Objective:

To see if the antidepressant response of ketamine is linked to AMPA receptors.

Eligibility:

Adults ages 18-70 with major depression disorder without psychotic features

Design:

Participants will be screened under protocol 01-M-0254. They will have blood tests and a physical exam.

Participants will stay at the NIH Clinical Center for 5 weeks.

Phase 1 lasts 4 weeks. For 2 weeks, participants will taper off their psychiatric medicine. Then they will have the following tests:

* Blood draws
* Psychological tests
* MRI: Participants will lie in a machine that takes pictures of their brain.
* MEG: Participants will lie down and do tasks. A cone lowered on their head will record brain activity.
* Optional sleep tests: Electrodes on the scalp and body and belts around the body will monitor participants while they sleep.
* Optional TMS: Participants will do tasks while a wire coil is held on their scalp. An electrical current will pass through the coil that affects brain activity.

For phase 2, on day 0 participants will take the study drug or a placebo orally. While having a MEG, they will get ketamine infused into a vein in one arm while blood is drawn from a vein in the other arm. On day 1, participants will again take the study drug or a placebo orally. On days 3-7, they will repeat many of the phase 1 tests. Days 8 and 9 are optional and include an open label ketamine treatment and many of the phase 1 tests.

DETAILED DESCRIPTION:
Objective

Work by our group and others has demonstrated that a single intravenous dose of the glutamatergic modulator ketamine consistently produces rapid (within two hours), robust, and relatively sustained (approximately one to two weeks) antidepressant effects in patients with treatment-resistant major depressive disorder (MDD) and bipolar depression. Although ketamine is an N-methyl-D-aspartate (NMDA) receptor (NMDAR) antagonist, convergent evidence from behavioral, cellular, and molecular ketamine studies supports the theory that enhanced -amino-3-hydroxy-5-methyl-4-isoxazolepropionic acid (AMPA) receptor activity-with a concomitant increase in synaptic plasticity-is critical to its mechanism of antidepressant action and may be the key to developing analogous rapidacting antidepressants. Notably, both animal and human studies indicate that acute, sub-anesthetic ketamine infusion is associated with robust increases in gamma power. Multiple synaptic mechanisms play a role in regulating gamma oscillations, including AMPA receptor (AMPAR)-mediated depolarization and gamma aminobutyric acid (GABA) receptor-mediated inhibition. Ketamine may influence both of these systems, both by silencing GABAergic inhibitory synapses and by increasing glutamate release, thereby activating AMPARs.

This clinical translational mechanistic protocol, in parallel with a preclinical study (Bench-to-Bedside Award, NIH), is designed to begin to disentangle the neurobiological underpinnings of ketamine s mechanism of antidepressant action and to develop a cross-species biomarker of target engagement (i.e., gamma power). The study will test the importance of AMPAR throughput by attempting to block the behavioral (i.e., antidepressant), electrophysiological, and biochemical effects of ketamine with an AMPAR antagonist. We first demonstrated in animal models that administering an AMPAR antagonist (NBQX) could block ketamine s antidepressant-like properties, suggesting that AMPAR neurotransmission was involved in these effects. This finding has now been replicated by multiple labs. In the present study, we propose to evaluate whether pre-treatment with perampanel, an AMPAR antagonist, blocks or reduces the acute antidepressant effects of ketamine in patients with treatment resistant depression (TRD). Further, we will examine whether AMPAR activity is important to the continued antidepressant effects of ketamine by examining whether treatment with perampanel blocks or reduces ketamine s continued antidepressant effects.

Study Population

70 patients ages 18 to 70 years, with a diagnosis of MDD (without psychotic features) will be recruited for this study.

Study Design

This is a two-phase pathophysiological study that attempts to understand the mechanism of action of ketamine s antidepressant effects. Phase I includes a medication taper, drug-free period, and baseline testing (e.g. clinical rating scales, sEEG, TMS, MEG). In Phase II, participants will receive an open-label ketamine infusion with a randomized, double-blind, add-on intervention (perampanel vs. placebo). Two to three hours prior to receiving ketamine (0.5 mg/kg), subjects will be randomized into one of three arms. Subjects in Arm 1 will receive perampanel (8 mg p.o.), while those randomized to Arm 2 or Arm 3 will receive matching placebo. On Day 1, the second blinded oral medication will be administered after clinical rating scales are obtained. Subjects randomized to Arm 1 and 3 will receive matching placebo, while subjects randomized to Arm 2 will receive perampanel. sEEG, TMS, and MEG will be obtained again on two more occasions during Phase II. Participants who completed Phase II will also be offered one open-label ketamine treatment, during which they will be assessed for mood symptoms and possible side effects.

Outcome Measures

The primary outcome measure is the Montgomery-Asberg Depression Rating Scale (MADRS). Hypothesis 1: By Day 1, patients treated with ketamine who are randomized to pre-treatment with a single oral dose of the AMPAR antagonist perampanel will have significantly more depressive symptoms than those who are randomized to pretreatment with placebo, as measured by the MADRS. Hypothesis 2: By Day 2, patients treated with ketamine who were randomized to perampanel on Day 1 will have significantly more depressive symptoms than those who were randomized to placebo, as measured by the MADRS. To acquire data corroborating that ketamine s antidepressant effects are mediated through AMPARs, surrogate plasticity measures will be obtained using sEEG, TMS, and MEG. In addition, blood samples for biomarkers will also be obtained.

ELIGIBILITY:
* INCLUSION CRITERIA:

Phases I-II

1. 18 to 70 years of age.
2. Each subject must have a level of understanding sufficient to agree to all required tests and examinations and sign an informed consent document.
3. All subjects must have undergone a screening assessment under protocol 01-M-0254, "The Evaluation of Patients with Mood and Anxiety Disorders and Healthy Volunteers".
4. Subjects must fulfill DSM-IV or -5criteria for Major Depression (Major Depressive Disorder) without psychotic features, based on clinical assessment and informed by a structured diagnostic interview (SCID-P).
5. Subjects must have an initial score on the MADRS greater than or equal to 22 and a YMRS score of <12 within one week of study entry and upon entry into Phase II.
6. Lack of response to two adequate antidepressant trials, with [at least] one in the current major depressive episode, operationally defined using the Antidepressant Treatment History Form (ATHF); a failed adequate trial of ECT [or TMS] would count as an adequate antidepressant trial.
7. Current major depressive episode lasting at least four weeks
8. Agree to be hospitalized

Open-Label Ketamine Treatment

1. Participants must have met all inclusion criteria for and completed Study Phase II
2. Individuals who are able to get pregnant must be willing to remain sexually abstinent or use at least one form of effective birth control during participation in Phase III.

EXCLUSION CRITERIA:

Phases I-II

1. Current psychotic features or a diagnosis of schizophrenia or any other psychotic disorder as defined in the DSM-IV or DSM-5.
2. Subjects with a history of substance abuse or dependence diagnosis (DSM-IV) or substance use disorder (DSM-5 equivalent) (except for caffeine or nicotine dependence) within the preceding 3 months. In addition, subjects who currently are using drugs (except for caffeine or nicotine) must not have used illicit substances or known drugs of abuse in the 2 weeks prior to screening and must have a negative alcohol and drug urine test (except for prescribed benzodiazepines or stimulants) at screening.
3. Serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease, coronary artery disease, atherosclerotic ischemic stroke, and atrial fibrillation), endocrinologic, neurologic, immunologic, or hematologic disease.
4. Pregnant or nursing individuals or those who are physically able to become pregnant. Participants who are physically able to become pregnant or cause a pregnancy must use at least one form of effective birth control or remain completely abstinent from sexual intercourse during the entire period of study participation (or until the last clinical labs and ratings). Participants able to become pregnant must have negative urine pregnancy tests no more than 24 hours prior to receiving the study drugs and undergoing imaging procedures.
5. Subjects with one or more seizures without a clear and resolved etiology or current use of medication known to lower seizure threshold. History of seizure (regardless of age or etiology), history of epilepsy in self or first-degree relatives, stroke, brain surgery, head injury, or known structural brain lesion will be excluded from the TMS procedures.
6. Presence of any medical illness likely to alter brain morphology and/or physiology (e.g., hypertension, diabetes) even if controlled by medications.
7. Clinically significant abnormal laboratory tests.
8. (For imaging procedures) Subjects with hearing loss that has been clinically evaluated and diagnosed and may be worsened through participation in imaging procedures
9. Positive HIV test
10. Weight > 119 kg
11. Treatment with any concomitant psychiatric medication prior to entering Phase II. [Medications must be tapered during Phase I.]
12. Treatment with any non-psychiatric medication/s.
13. Any use of opioid medication in the past 3 months
14. Treatment with a reversible monoamine oxidase inhibitor (MAOI) prior to entering Phase II. [Medications must be tapered during Phase I.]
15. Treatment with fluoxetine or aripiprazole at the time of screening.
16. Unwilling to stop undergoing structured, individualized psychotherapy. (Such therapy, including CBT, will not be permitted during Phases I and II of the study.)
17. Presence of metallic (ferromagnetic) implants (e.g., heart pacemaker, aneurysm clip).
18. Participants who are uncomfortable in small closed spaces (have claustrophobia).
19. Are unable to lie comfortably supine for up to 90 minutes and would feel uncomfortable in the MRI and MEG machines.
20. Subjects who, in the investigator s judgment, pose a current serious suicidal or homicidal risk.
21. Subjects who have a history of aggressive behavior towards others
22. A current NIMH employee/staff or their immediate family member

Open-Label Ketamine Treatment

1. Intolerable or serious adverse reaction to ketamine during Phase II
2. Participants with a positive urine for an illicit substance no more than 24 hours prior to ketamine treatment.
3. Pregnant or nursing individuals or those who plan to become pregnant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-01-21 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Acute Antidepressant Efficacy: Change from baseline Montgomery Asberg Depression Rating Scale (MADRS) score post ketamine infusion | Baseline, Day 1
  Clinical rating scale of depression
Continued Antidepressant Efficacy: Change from baseline MADRS score post treatment with ketamine with perampanel versus placebo. | Baseline, Day 1, Day 2 Day 7
  Clinical rating scale of depression

SECONDARY OUTCOMES:
Acute Antidepressant Efficacy: Change in slow wave activity/slope post ketamine infusion | Baseline (night), Day 1 (night)
  Polysomnography (PSG)/Electroencephalography (EEG) data
Acute Antidepressant Efficacy: Change in synaptic plasticity post ketamine infusion | Baseline, Day 1
  Transcranial Magnetic Stimulation (TMS) data
Continued Antidepressant Efficacy: Gamma power change from baseline post treatment with ketamine with perampanel versus placebo | Baseline, Day 1
  Magnetoencephalography (MEG) data
Continued Antidepressant Efficacy: Change in slow wave activity/slope from baseline post treatment with ketamine with perampanel versus placebo | Baseline (night), Day 1 (night)
  PSG/EEG data
Continued Antidepressant Efficacy: Change in synaptic plasticity from baseline post treatment with ketamine with perampanel versus placebo | Baseline, Day 1
  TMS data
Acute Antidepressant Efficacy: Gamma power change from baseline post ketamine infusion | Baseline, Day 1
  Magnetoencephalography (MEG) data
Acute Antidepressant Efficacy: Change in peripheral measures associated with the administration of ketamine | Baseline, Day 1, Day 2, Day 7
  Plasma/serum biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Zarate, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Clinical and demographic and biomarker participant data collected during the trial, after deidentification.
Supporting Information: SAP
Time Frame: Starting within 1 year of completion of the study.
Access Criteria: The Branch Chief will review requests and access will need to be approved by the NIMH/DIRP SD and OCD NIMH and the NIH IIRB.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-M-0107.html